CLINICAL TRIAL: NCT03098680
Title: A Study of the Pharmacokinetic and Pharmacodynamic Responses in Healthy and Altered Human Cardiovascular Systems
Acronym: PRIME
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit in time before end of PhD studentship
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Joseph Cheriyan, MD, Dr, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PRIME (A094136)
Record Dates: First submitted 2017-03-14; First posted 2017-04-04 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Drug-Related Side Effects and Adverse Reactions; Cardiovascular System Disease
Keywords: Adverse reactions; Cardiovascular; Translation; Modelling; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Cardiovascular Diseases | interventions — Albuterol; Nicardipine; Dobutamine; Phenylephrine; Verapamil; Phentolamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo, Salbutamol, Nicardipine, Dobutamine) (Experimental): Participants will receive each drug, to be given on separate study days. The drugs will be given as a 3 stage infusion with dose increasing at each stage. Each stage will be 30 minutes in duration.
  Placebo; Salbutamol(Albuterol) Sulfate (Dose: 2mcg/min, 5mcg/min, 10mcg/min); Nicardipine Hydrochloride (Dose: 1mg/hr, 2.5mg/hr, 5mg/hr); Dobutamine Hydrochloride (Dose: 1mcg/kg/min, 2.5mcg/kg/min, 5mcg/kg/min)
  Interventions: Drug: Albuterol Sulfate; Drug: Nicardipine Hydrochloride; Drug: Dobutamine Hydrochloride; Drug: Placebo
- Group B (Placebo, Phenylephrine, Verapamil, Phentolamine) (Experimental): Participants will receive each drug, to be given on separate study days. The drugs will be given as a 3 stage bolus with dose increasing at each stage. Each stage will be 30 minutes apart.
  Placebo; Phenylephrine Hydrochloride (Dose: 100mcg, 200mcg, 300mcg); Verapamil Hydrochloride (Dose: 1mg, 2.5mg, 5mg); Phentolamine Mesylate (Dose: 1mg, 2mg, 3mg)
  Interventions: Drug: Phenylephrine Hydrochloride; Drug: Verapamil Hydrochloride; Drug: Phentolamine Mesylate; Drug: Placebo

INTERVENTIONS:
Drug: Albuterol Sulfate — see arm/group descriptions
  Other Names: Salbutamol Sulfate
  Arms: Group A (Placebo, Salbutamol, Nicardipine, Dobutamine)
Drug: Nicardipine Hydrochloride — see arm/group descriptions
  Arms: Group A (Placebo, Salbutamol, Nicardipine, Dobutamine)
Drug: Dobutamine Hydrochloride — see arm/group descriptions
  Arms: Group A (Placebo, Salbutamol, Nicardipine, Dobutamine)
Drug: Phenylephrine Hydrochloride — see arm/group descriptions
  Arms: Group B (Placebo, Phenylephrine, Verapamil, Phentolamine)
Drug: Verapamil Hydrochloride — see arm/group descriptions
  Other Names: Securon IV
  Arms: Group B (Placebo, Phenylephrine, Verapamil, Phentolamine)
Drug: Phentolamine Mesylate — see arm/group descriptions
  Other Names: Phentolamine Mesilate
  Arms: Group B (Placebo, Phenylephrine, Verapamil, Phentolamine)
Drug: Placebo — see arm/group descriptions
  Other Names: 0.9% Sodium Chloride

SUMMARY:
Unwanted effects on the cardiovascular system is one of the most common causes of safety related discontinuation of a drug. This study aims to develop an in silico model of the human cardiovascular system that can be used to predict unwanted cardiovascular effects of drugs. This will be achieved through a drug administration study that will generate comprehensive pharmacokinetic and pharmacodynamic data following the administration of the following drugs, all known to have effects on the cardiovascular system. Half the participants will receive: Placebo, Salbutamol, Nicardipine, Dobutamine and the other half will receive Placebo, Phenylephrine, Verapamil, Phentolamine.

DETAILED DESCRIPTION:
Safety is an integral part of developing new medicines. Potential drugs can be withdrawn from development at any stage of the process if there are concerns over safety. In recent years, computer models that recreate physiology have been increasingly adopted in various aspects of drug development, including safety, to predict the effects of new drugs. The accuracy of this predictive model is however, dependent on the ability for animal data (which the model is usually based on) to be 'translated' to human data. As no animal is identical to humans, the difference between species needs to be understood for the model to be accurate.

Unwanted effects on the cardiovascular system is one of the most common causes of safety related discontinuation of a drug. The present study focuses on generating high quality human cardiovascular data that is comparable with existing animal data. This will be achieved through the collection of detailed pharmacokinetic and pharmacodynamic data following administration of drugs that are known to affect the cardiovascular system through a range of mechanisms. This will be first performed in healthy participants before extending it to those with pre-existing (or risk-factors for) cardiovascular disease. The aim is to understand the differences between species and the study populations and using the collected data to help inform how a translational model is to be built.

Study Design: Single centre, single (participant) blind, within subject, drug administration study

Drugs used in study:

1. Salbutamol - a beta-2-adrenergic agonist
2. Nicardipine - a dihydropyridine calcium channel antagonist
3. Dobutamine - a beta-1-adrenergic agonist
4. Phenylephrine - a selective alpha-1-adrenergic agonist
5. Verapamil - a phenylalkylamine calcium channel antagonist
6. Phentolamine - a non-selective alpha adrenergic antagonist

Study Population:

The study will take place in three parts (A, B and C), with each part representing population groups that are of interest.

Part A (16 participants): Healthy individuals with no identifiable cardiovascular risk factors will be recruited for this part of the study. The aim of this part is to enable the collection of physiological data after drug administration in a 'normal' cardiovascular system.

Part B (8 participants): Part B will involve the recruitment of participants who may possess an altered/challenged cardiovascular system. Participants recruited will possess one of the following factors: known diagnosis of diabetes, known diagnosis of hypertension, obesity (BMI>30), age >65. The data collected will provide information on how potential changes to baseline cardiovascular physiology may affect the effect of the drug.

Part C (8 participants): In order to understand the impact of medicines on cardiovascular physiology in the absence of the autonomic nervous system regulation, we will recruit participants with dysfunction of the autonomic system to Part C of the study.

Maximum duration of participation for each participant:

1x screening (1 hour duration), 4x study visits (8 hour duration each) with minimum 72 hours gap in between visits. Maximum duration is 4 months to complete all visits.

ELIGIBILITY:
Part A Inclusion Criteria

To be included in the study the patient must:

* Have given written informed consent to participate
* Male
* Be aged between 18 and 30 years at the time of first study appointment
* BMI <30
* Deemed healthy to partake in the study at the discretion of the investigator

Exclusion Criteria

The presence of any of the following will preclude patient inclusion:

* Less than 18 years old, >30 years old
* BMI >30
* On regular medications
* Known allergy to medications
* History of psychiatric, chronic cardiac / respiratory / renal disease
* Known diagnosis of diabetes
* Habitual smoker
* Screening heart rate of less than 60 beats per minute
* Screening heart rate of greater than 100 beats per minute
* Screening blood pressure of less than 100mmHg systolic and/or 55mmHg diastolic
* Any concomitant condition or circumstance that, at the discretion of the investigator, may affect the participant's ability to complete the study
* Current participation in another interventional research study

Part B Inclusion Criteria

To be included in the study the patient must:

* Have given written informed consent to participate
* Male
* Be aged over 18 years at the time of first study appointment
* Possess one of the following - known diagnosis of diabetes, known diagnosis of hypertension, obesity (BMI>30), aged >65
* Deemed healthy to partake in the study at the discretion of the investigator

Exclusion Criteria

The presence of any of the following will preclude patient inclusion:

* Less than 18 years old
* On regular medications that are contraindicated for co-use with the study drugs
* Known allergy to medications
* Screening heart rate of less than 60 beats per minute
* Screening heart rate of greater than 100 beats per minute
* Screening blood pressure of less than 100mmHg systolic and/or 55mmHg diastolic
* Any concomitant condition or circumstance that, at the discretion of the investigator, may affect the participant's ability to complete the study
* Current participation in another interventional research study

Part C Inclusion Criteria

To be included in the study the patient must:

* Have given written informed consent to participate
* Male
* Be aged over 18 years at the time of first study appointment
* Clinical diagnosis of autonomic dysfunction
* BMI<30
* Deemed healthy to partake in the study at the discretion of the investigator

Exclusion Criteria

The presence of any of the following will preclude patient inclusion:

* Less than 18 years old
* BMI >30
* On regular medication
* Known allergy to medications
* History of psychiatric, chronic cardiac / respiratory / renal disease
* Habitual smoker
* Screening heart rate of less than 60 beats per minute
* Screening heart rate of greater than 100 beats per minute
* Screening blood pressure of less than 100mmHg systolic and/or 55mmHg diastolic
* Any concomitant condition or circumstance that, at the discretion of the investigator, may affect the participant's ability to complete the study
* Current participation in another interventional research study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Heart rate | At every study visit (each lasting up to 8 hours)
  Change in heart rate from baseline over time after administration of drug
Peripheral blood pressure | At every study visit (each lasting up to 8 hours)
  Change in resting peripheral blood pressure (systolic, diastolic, pulse pressure and mean pressure) over time after administration of drug
Central blood pressure | At every study visit (each lasting up to 8 hours)
  Change in resting central aortic pressure (systolic, diastolic, pulse pressure and mean pressure) from baseline over time after administration of drug
Cardiac output | At every study visit (each lasting up to 8 hours)
  Change in cardiac output from baseline over time after administration of drug
Stroke volume | At every study visit (each lasting up to 8 hours)
  Change in stroke volume from baseline over time after administration of drug
ECG/Cardiac monitor | At every study visit (each lasting up to 8 hours)
  Change in ECG (PR interval/QRS interval/QT interval/QTc interval/RR interval) over time after administration of drug

SECONDARY OUTCOMES:
Plasma drug concentration (all drugs) | These will be measured during each part of the study, estimated 6 months per part. Taken at: -(5mins, 10mins,15mins, 30mins, 35mins, 40mins, 45mins, 60mins, 65mins, 70mins, 75mins, 90mins, 120mins, 150mins, 180mins, 240mins, 360mins)
  Measure of drug levels (parent compound and active metabolites) at the specified time points
Plasma drug (active) metabolite concentration (varapamil only) | Throughout the study, estimated 6 months per part. Taken at specified timepoints (5mins, 10min, 15mins, 30mins, 35mins, 40mins, 45mins, 60mins, 65mins, 70mins, 75mins, 90mins, 120mins, 150mins, 180mins, 240mins, 360mins)
  Measure of drug levels (parent compound and active metabolites) at the specified time points
Renal Function | Through study completion, up to 4 months
  Changes in renal function throughout study
Liver function | Through study completion, up to 4 months
  Changes in liver function throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MBCHB, MA, FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No